CLINICAL TRIAL: NCT02037217
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Thalamotomy in the Treatment of Essential Tremor
Brief Title: ExAblate Transcranial MR Guided Focused Ultrasound in the Treatment of Essential Tremor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET001K
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExAblate Treatment (Experimental)
  Interventions: Device: ExAblate Transcranial MRgFUS System

INTERVENTIONS:
Device: ExAblate Transcranial MRgFUS System

SUMMARY:
A feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MRI-guided focused ultrasound (MRgFUS) treatment of patients with medication-refractory movement disorders, namely Essential Tremor (ET).

This study is designed as a prospective, single site, single arm, nonrandomized study. Assessments will be made before and three months after MRgFUS for clinical symptom relief, quality of life (QoL) improvements, and safety of MRgFUS in the treatment of ET. Similarly, QoL measures will be obtained using Quality of Life in Essential Tremor (QUEST) questionnaire. Relative Safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study. This study will be performed on the 3T MR scanners.

The ExAblate system is a medical device that involves a focused ultrasound system and an MRI scanner. ExAblate delivers a pulse of focused ultrasound energy, or sonication, to the targeted tissue. In this particular study the targeted tissue is a unilateral thermal lesion created in the ventralis intermedius nucleus of the thalamus.

The treatment begins with a series of standard diagnostic MR images to identify the location and shape of tumor to be treated. The ExAblate computer uses the physician's designation of the target volume to plan the best way to cover the target volume with small spots called "sonications". These treatment spots are cylinder shaped. Their size depends on sonication power and duration. During the treatment, a specific MR scan, which can be processed to identify changes in tissue temperature, provides a thermal map of the treatment volume to confirm the therapeutic effect. The thermal map is used to monitor the treatment in progress, and confirm that the ablation is proceeding according to plan, thus closing the therapy loop.

The ExAblate transcranial operates a helmet-shaped transducer (currently utilizing 1000-element phased array transducer) positioned above the subject head. The ExAblate transcranial system also includes means to immobilize the subject head, cool the interface water, and software for CT analysis and phase correction computation.

The ExAblate transcranial system is an experimental device and is being investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between 18 and 80 years, inclusive
2. Patients who are able and willing to give consent and able to attend all study visits
3. A diagnosis of ET as confirmed from clinical history and examination by a movement disorder neurologist
4. Tremor refractory to adequate trials of at least two medications, one of which should be either propranolol or primidone. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
5. Vim nucleus of thalamus can be target by the ExAblate device. The Vim region of the thalamus must be apparent on MRI such that targeting can be performed with either direct visualization or by measurement from a line connecting the anterior and posterior commissures of the brain.
6. Able to communicate sensations during the ExAblate MRgFUS treatment
7. Postural or intention tremor severity score of greater than or equal to 2 in the dominant hand/arm as measured by the CRST rating scale.
8. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
9. May have bilateral appendicular tremor
10. Significant disability due to essential tremor despite medical treatment (CRST score of 2 or above in any one of the items 16-23 from the Disability subsection of the CRST: [speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities])
11. Inclusion and exclusion criteria have been agreed upon by two members of the medical team.

Exclusion Criteria:

1. Patients with unstable cardiac status including:

   1.1 Unstable angina pectoris on medication 1.2 Patients with documented myocardial infarction within six months of protocol entry 1.3 Congestive heart failure requiring medication (other than diuretic) 1.4 Patients on anti-arrhythmic drugs
2. Patients exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:

   * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
   * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
3. Severe hypertension (diastolic BP > 100 on medication)
4. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
5. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
6. Severely impaired renal function (estimated glomerular filtration rate < 45ml/min/1.73 m2) or receiving dialysis
7. History of abnormal bleeding and/or coagulopathy
8. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
9. Active or suspected acute or chronic uncontrolled infection
10. History of intracranial hemorrhage
11. Cerebrovascular disease (multiple CVA or CVA within 6 months)
12. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
13. Symptoms and signs of increased intracranial pressue (e.g. headache, nausea, vomiting, lethargy, and papilledema)
14. Are participating or have participated in another clinical trial in the last 30 days
15. Patients unable to communicate with the investigator and staff.
16. Presence of any other neurodegenerative disease like parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer"s disease.
17. Anyone suspected to have the diagnosis of idiopathic Parkinson"s disease. This includes excluding anyone with the presence of parkinsonian features including bradykinesia rigidity, or postural instability. Subjects who exhibit only mild resting tremor but no other symptoms or signs of PD may be included.
18. Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
19. History of immunocompromise, including patient who is HIV positive
20. Known life-threatening systemic disease
21. Patients with a history of seizures within the past year
22. Patients with current or a prior history of any psychiatric illness will be excluded. Any presence or history of psychosis will be excluded. Patients with mood disorders including depression will be excluded. For the purpose of this study, we consider a significant mood disorder to include any patient who has:

    * been under the care of a psychiatrist for over 3 months
    * taken antidepressant medications for greater than 6 months
    * has participated in cognitive-behavioral therapy
    * been hospitalized for the treatment of a psychiatric illness
    * received transcranial magnetic stimulation
    * received electroconvulsive therapy
23. Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy
24. Patients with brain tumors
25. Any illness that in the investigator's opinion preclude participation in this study.
26. Pregnancy or lactation.
27. Legal incapacity or limited legal capacity.
28. Patients who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Device or procedure related Adverse Events reported | 3 Months
  Safety of the ExAblate transcranial treatment will be determined by an evaluation of the incidence and severity of device and procedure related complications from the first / treatment day visit through the 3-Months post-treatment time point. All AEs will be reported and categorized by investigators as definitely, probably, possibly, or unrelated to the device, procedure, or post-surgical changes in neurological status. Alternative treatments resulting from post-surgical changes in neurological status will be reported.

SECONDARY OUTCOMES:
Tremor rating scales: the Clinical Rating Scale for Tremors | 3 Month
  Primary effectiveness will be evaluated using validated, tremor rating scales: the Clinical Rating Scale for Tremors (CRST) for ET patients, based upon patients in whom unilateral ExAblate lesioning is attempted (i.e., Intent-to-Treat analysis). Efficacy is defined as a reduction in contralateral symptoms at 3-months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Chang, Prof., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- See also: Sponsor website — http://www.insightec.com